CLINICAL TRIAL: NCT07256678
Title: Jewel P-WCD Post-Approval Study (PAS)
Status: Not yet recruiting | Type: Observational
Sponsor: Element Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-3162
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Jewel-P WCD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This study is an observational registry study of the Jewel P-WCD in post-market use
  Interventions: Other: This study is an observational registry study of the Jewel P-WCD in post-market use; Other: Jewel

INTERVENTIONS:
Other: This study is an observational registry study of the Jewel P-WCD in post-market use — This study is an observational registry study of the Jewel P-WCD in post-market use
Other: Jewel — This study is an observational registry study of the Jewel P-WCD in post-market use

SUMMARY:
The objective of this PAS is to demonstrate the continued safety and clinical effectiveness of the Jewel P-WCD.

DETAILED DESCRIPTION:
This study is an observational registry study of the Jewel P-WCD in post-market use

ELIGIBILITY:
Inclusion Criteria:

* N/A - registry will collect data already obtained commercially from patients prescribed the Jewel P-WCD.

Exclusion Criteria:

* N/A - registry will collect data already obtained through commercial consent from patients prescribed the Jewel P-WCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population who are at elevated risk of Sudden Cardiac Arrest (SAC) while they wait for permanent diagnosis.
Sampling Method: Probability Sample
Enrollment: 6330 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percent of VT/VF events successfully detected by the Jewel P-WCD | From enrollment to the end of treatment at approximately 90 days

IPD SHARING:
Plan to Share IPD: No